CLINICAL TRIAL: NCT03995069
Title: Novel Training Environment to Normalize Altered Finger Force Direction Post Stroke
Acronym: NEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3066-R; NCT03993756 (obsolete NCT alias)
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: Hand Strength; Electromyography
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D (Experimental): The participant's voluntary grip forces in all 3 dimensions will be shown to the participant via computer screen.
  Interventions: Behavioral: 3D
- 1D (Active Comparator): The participant's voluntary grip force in 1 dimension will be shown to the participant via computer screen.
  Interventions: Behavioral: 1D

INTERVENTIONS:
Behavioral: 3D — Practice generating grip force to the target shown on the computer screen in 3 dimensions.
  Arms: 3D
Behavioral: 1D — Practice generating grip force to the target shown on the computer screen in 1 dimension.
  Arms: 1D

SUMMARY:
Despite the functional importance, fingertip forces are rarely explicitly addressed with feedback in therapy. This gap in treatment is due to a lack of tools to provide explicit feedback on patients' volitional finger force generation. To address this unmet need, the investigators developed a novel tool for practice of volitional three-dimensional (3D) force generation with explicit feedback. The objective of this project is to determine if 3D finger force training is an effective tool in restoring hand function post stroke.

DETAILED DESCRIPTION:
Despite the functional importance, fingertip forces are rarely explicitly addressed with feedback in therapy. This gap in treatment is due to a lack of tools to provide explicit feedback on patients' volitional finger force generation. To address this unmet need, the investigators developed a novel tool for practice of volitional three-dimensional (3D) force generation with explicit feedback. The objective of this project is to determine if 3D finger force training is an effective tool in restoring hand function post stroke.

Stroke survivors with moderate to severe hand impairment with at least palpable volitional grip force will randomly be assigned to either the experimental or control group, stratified by impairment level. Both groups will undergo 3 1-hr training sessions per week for 6 weeks in which they practice volitional finger force generation against force sensors. The experimental group will practice for various target force directions to explore the 3D force workspace and receive feedback in 3D force, while the control group will practice 1D force generation without feedback on other directional forces on a computer screen.

Training will progress by increasing influence of flexion synergy by varying posture requirements and increasing force level, introducing feedback delay, and incorporating unilateral/bilateral activity. Evaluation will occur at baseline (3 times over 3 weeks to establish baseline trends) and every 2 weeks during 6-week intervention to determine pattern of progress, and at 1-month follow-up to assess retention.

ELIGIBILITY:
Inclusion Criteria:

* Survived a stroke at least 3 months ago
* Moderate to severe hand impairment (Chedoke-McMaster Hand Stage 2-4)
* Ability to generate palpable volitional grip force upon cue
* Sufficient cognitive ability to participate (NIH Stroke Scale, NIHSS, Questions and Commands score = 0-1)
* Ability to recognize all quadrants of the visual field (NIHSS Visual Field Test score = 0)

Exclusion Criteria:

* Concurrent upper limb rehabilitation
* Inability to follow 2-step commands
* Severe muscle tone prohibiting passive movement of the fingers or proper placement of the fingers on the force sensors as needed to participate in the training (Modified Ashworth Scale=4-5 out of 5)
* Change in spasticity medication or botulinum toxin injection in the upper limb within 3 months prior to or during enrollment
* Total sensory loss on fingertips (NIHSS Sensory score=2)
* Comorbidity (e.g., orthopaedic conditions that limit ranges of motion, premorbid neurologic conditions)
* Language barrier or cognitive impairment that precludes providing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Na Jin Seo, PhD MS BS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data will be shared as a supplement of a publication in peer reviewed journals if allowed by the journal, and also upon written request.
Supporting Information: Study Protocol
Time Frame: During the study period and 5 years post study completion

REFERENCES:
- [Derived] Seo NJ, Schranz C, Coupland K, Blaschke J, Scronce G, Finetto C, Baker A, Gallant J, Alston A, Howard K, Thompson D, Ramakrishnan V, Holmstedt CA, Kamper DG. Biofeedback Training for 3-Dimensional Finger Force Control to Improve Upper Limb Function Poststroke: An RCT. Stroke. 2025 Aug;56(8):2266-2276. doi: 10.1161/STROKEAHA.125.050965. Epub 2025 May 22. PMID 40401398
- [Derived] Seo NJ, Kamper DG, Ramakrishnan V, Harvey JB, Finetto C, Schranz C, Scronce G, Coupland K, Howard K, Blaschke J, Baker A, Meinzer C, Velozo CA, Adams RJ. Effect of novel training to normalize altered finger force direction post-stroke: study protocol for a double-blind randomized controlled trial. Trials. 2022 Apr 12;23(1):301. doi: 10.1186/s13063-022-06224-w. PMID 35413931

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Not meeting inclusion criteria (n=1) Declined to participate (n=3) Funding ended (n=2)
Groups:
- Visual Feedback of 3D Digit Force: The participant's voluntary grip forces in all 3 dimensions will be shown to the participant via computer screen.
  3D: Practice generating grip force to the target shown on the computer screen in 3 dimensions.
- Visual Feedback of 1D Digit Force: The participant's voluntary grip force in 1 dimension will be shown to the participant via computer screen.
  1D: Practice generating grip force to the target shown on the computer screen in 1 dimension.
Period: Overall Study
Arm/Group | Visual Feedback of 3D Digit Force | Visual Feedback of 1D Digit Force
Started | 22 | 23
Completed | 16 | 17
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Visual Feedback of 3D Digit Force | Visual Feedback of 1D Digit Force | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12) | 60 (9) | 59 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 13 | 14 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Action Research Arm Test (ARAT)
Description: change in a clinical assessment, ARAT, that is in a scale 0-57 with a higher score representing better upper extremity function
Time Frame: baseline to within 1 week post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Visual Feedback of 3D Digit Force | Visual Feedback of 1D Digit Force
Number analyzed (Participants) | 17 | 19
score on a scale | 3.5 (0.65) | 0.8 (0.66)

2. Other Pre Specified Outcome: Box and Block Test
Description: a clinical assessment measuring the number of blocks that a person can move in a minute, with a higher score representing better upper extremity function
Time Frame: baseline to within 1 week post intervention
Measure: Mean (Standard Error); unit: blocks moved in 1 min
Arm/Group | Visual Feedback of 3D Digit Force | Visual Feedback of 1D Digit Force
Number analyzed (Participants) | 17 | 19
blocks moved in 1 min | 3.03 (0.97) | 0.92 (0.95)

3. Other Pre Specified Outcome: Stroke Impact Scale Hand Subscale
Description: Perceived difficulty in using the affected hand for activities of daily living. Scale 0-100. A higher score represents better function (less difficulty).
Time Frame: baseline to within 1 week post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Visual Feedback of 3D Digit Force | Visual Feedback of 1D Digit Force
Number analyzed (Participants) | 17 | 19
score on a scale | 12 (2) | 6 (2)

4. Other Pre Specified Outcome: Action Research Arm Test
Description: change in a clinical assessment of Action Research Arm Test that is in a scale 0-57 with a higher score representing better upper extremity function
Time Frame: baseline to 1 month post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Visual Feedback of 3D Digit Force | Visual Feedback of 1D Digit Force
Number analyzed (Participants) | 16 | 17
score on a scale | 3.9 (0.7) | 0.7 (0.7)

5. Other Pre Specified Outcome: Box and Block Test
Description: a clinical assessment for upper extremity function.
Time Frame: baseline to 1 month post intervention
Measure: Mean (Standard Error); unit: blocks moved in 1 min
Arm/Group | Visual Feedback of 3D Digit Force | Visual Feedback of 1D Digit Force
Number analyzed (Participants) | 16 | 17
blocks moved in 1 min | 2.5 (1) | 0.5 (1)

6. Other Pre Specified Outcome: Stroke Impact Scale Hand Subscale
Description: as for outcome 3
Time Frame: baseline to 1 month post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Visual Feedback of 3D Digit Force | Visual Feedback of 1D Digit Force
Number analyzed (Participants) | 16 | 17
score on a scale | 15 (2) | 8 (2)

ADVERSE EVENTS:
Time Frame: During the study participation (approximately 10 weeks)
Arm/Group | Visual Feedback of 3D Digit Force | Visual Feedback of 1D Digit Force
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/22 | 3/23
Other Adverse Events (participants affected / at risk) | 18/22 | 18/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Visual Feedback of 3D Digit Force (N=22) | Visual Feedback of 1D Digit Force (N=23)
drug abuse (General disorders) | 1 | 0
tremor with new seizure medication (Nervous system disorders) | 1 | 0
car accident (General disorders) | 0 | 1
transient amnesia, blackout (General disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Visual Feedback of 3D Digit Force (N=22) | Visual Feedback of 1D Digit Force (N=23)
other adverse events (General disorders) | 18 | 18 — high blood pressure, dog bite, sore throat, fatigue, pain, etc.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT03995069/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT03995069/ICF_002.pdf